CLINICAL TRIAL: NCT00919386
Title: Three Methods of Ureteral Stent Measurement: Which Method Improves Quality of Life After Ureteral Stenting?
Brief Title: Ureteral Stent Size Measurement Study
Status: Completed | Type: Observational
Sponsor: CAMC Health System (Other)
Responsible Party: Principal Investigator, Samuel Deem, DO, Dr. Samuel Deem, CAMC medical Staff - With Admitting Privileges., CAMC Health System
Other Study IDs: 09-03-2137
Record Dates: First submitted 2009-05-15; First posted 2009-06-12 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Quality of Life
Keywords: Ureteric Measurement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1 Direct ureteric measurement: This is determined by using a 5 French Pollack Open-Ended Flexi-Tip Ureteral catheter (Cook, Spencer, Indiana) to cannulate the ureteral orifice. A retrograde pyelogram will be done at the conclusion of the procedure and the Pollack will be advanced to the pyeloureteral junction (PUJ) under fluoroscopy. At this point the length of the distance between the PUJ and vesicoureteral junction (VUJ) will be recorded and stent length determined based on this measurement.
- 2 Based on patient height: We will use the height measurement criteria used by Lee et al in their study. Patients less than 5'2" will receive a 22 cm stent, 5'3"-5'7" will get a 24 cm stent, 5'8"-5'10" will get a 26 cm stent, 5'11" to 6'1" will get a 28 cm stent, and all patients greater than 6'2" will receive a 30 cm stent.
- 3 Based on a predetermined formula: We will use the formula described by Wieder. Stent length in cm= patients height in inches - 42.

SUMMARY:
To examine a patient's quality of life using three methods for measuring stent size: (a) direct measurement, (b) patient height, and (c) a standardized formula. The intent of the study is to show if there is a difference in a patient's quality of life, postoperative symptoms, pain medication and anticholinergic use by using one of these specific methods for stent size determination. No method is interventional in this study.

DETAILED DESCRIPTION:
Ureteral stent placement is common in Urologic practice and many studies have been done looking at factors to improve stent related symptoms, but few have used a validated questionnaire to assess these symptoms affect on quality of life.We plan to prospectively randomize patients to three separate techniques such as (a) direct measurement,(b) patient height, and (c) a standardized formula for the determination of stent size. Using a validated questionnaire, the Ureteral Stent Symptoms Questionnaire (USSQ), we will assess whether there is a difference in outcome measures such as patient quality of life, need for pain medications and anticholinergics, and in postoperative symptoms based on one of these techniques. The USSQ was developed by Joshi et al to assess the impact of health-related quality of life issues related to ureteral stents. Data from USSQ questionnaire will be collected 7-10 days post-operatively as well as 4 weeks post-op and then this will be aggregated for our outcome measures to determine which method of stent size give better outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting to Charleston Area Medical Center between the ages of 18 and 90 years old who will undergo cytoscopy or ureteroscopy with ureteral stent placement will be eligible for the study.

Exclusion Criteria:

* Patients excluded from this study will be those who are less than 18 years of age, pregnant women, and patients who are septic on presentation, as well as patients who have had lower extremity amputations or are wheelchair bound.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community patients who present to Charleston area Medical Center (CAMC) or the private urology clinics of Drs. Davalos,Martinez,Tierney with the requirement of ureteral stent would be screened for possible enrillment in the study.
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2009-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
To determine the difference in patient quality of life (QOL), post-op symptoms, and pain medication and anticholinergic use in patients who receive ureteral stents where size is determined by direct measurement, patient height,a standardized formula. | within 4 weeks post-porcedure

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Deem, M.D., Principal Investigator — CAMC Medical Staff - with admitting privileges
Locations (1):
- Urology center of charleston, Charleston, West Virginia, United States